CLINICAL TRIAL: NCT04760613
Title: A Phase I/II, Randomized, Double-blind, Placebo-controlled, Single-center Study of the Effects of Cannabidiol (CBD) on Opioid Plasma Levels in Participants With Chronic Radiculopathic Pain Syndromes Maintained on Chronic Opioid Therapy (COT)
Brief Title: CBD for Chronic Radicular Pain on Chronic Opioid Therapy (COT)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: s21-00230; 19-A0-00-1002274 (Other Grant/Funding Number: NIDA-CTN)
Record Dates: First submitted 2021-02-17; First posted 2021-02-18 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Radiculopathy
Keywords: Cannabidiol
MeSH Terms: conditions — Radiculopathy | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The trial will employ a double-blind pharmacologic intervention methodology where the investigational drug (CBD) and matched placebo oral pills will be masked in identically appearing capsules provided by the drug sponsor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (CBD) (Active Comparator)
  Interventions: Drug: Cannabidiol
- Placebo (PCB) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — 600 mg oral daily use (each capsule of active drug contains 50 mg of CBD)
  Arms: Cannabidiol (CBD)
Drug: Placebo — identical capsules containing placebo (taken daily by mouth)
  Arms: Placebo (PCB)

SUMMARY:
This double-blind, placebo-controlled, exploratory trial is designed to compare effects of oral CBD 600mg to placebo (PCB) in 20 outpatients with chronic spinal radiculopathies (without co-occurring Opioid Use Disorder), maintained on stable opioid analgesics for a minimum of 1 month. The trial duration will be approximately 2 weeks (from the point of randomization) of daily CBD 600mg vs placebo. Safety and tolerability of CBD will be assessed throughout the trial. The secondary efficacy outcome is change in pain outcomes from baseline to end of the treatment period at 2-weeks post-randomization/initiation of treatment with a Mixed Model for Repeated Measures (MMRM) statistical analysis performed to assess between group treatment effects of CBD relative to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥18
* Diagnosis of radicular CNCP (i.e. lumbar, cervical, thoracic)
* Maintained on stable dose opioid therapy for a minimum of 1 month

  o Note: Morphine Equivalent Daily Dose (MEDD) will be calculated using 2 reference documents: Guideline and conversion table to calculate MEDD from Centers for Medicaid and Medicare Services (CMS); Guidelines from the Centers for Disease Control and Prevention (CDC) intended for calculating total daily dose of opioids for safer dosage of opioid pharmacotherapy
* Able to provide voluntary informed consent
* If a woman of childbearing potential or a man, are willing to use approved form of contraception from screening for duration of the trial

Exclusion Criteria:

* Exclusionary medical conditions (e.g., unstable cardiac, hepatic, renal, neurologic illness) or any medical illness that in the opinion of the study physician poses a potential medical danger to the participant
* Exclusionary laboratory abnormalities (clinically significant abnormalities of complete blood count or chemistries, significantly impaired liver function)
* Current substance use disorder (including Opioid Use Disorder) other than nicotine or caffeine
* At screening, a positive urine toxicology test for: amphetamines (AMP), barbiturates (BAR), buprenorphine (BUP), benzodiazepines (BZO), cocaine (COC), 3,4-methylenedioxymethamphetamine (MDMA), methamphetamine (MET), methadone (MTD), phencyclidine (PCP), and tetrahydrocannabinol (THC)
* At screening, an alcohol level greater than 0 on a breathalyzer
* Severe psychiatric conditions including past or current DSM5 diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder
* Current significant suicidality (assessed using the C-SSRS), any suicidal behavior in the past 12 months, or any history of suicide attempts
* Current use of recreational or medical cannabis or any product containing CBD
* Pregnancy or lactation
* Current use of concomitant medications metabolized primarily by CYP2C19 isoenzymes
* Current use of concomitant medications significantly or primarily metabolized by CYP3A4 with the potential for adverse drug-drug interactions with CBD (i.e., ketoconazole, rifampicin)
* Current use of concomitant medications with a narrow therapeutic window significantly or primarily metabolized by CYP2C9 with the potential for adverse drug-drug interactions with CBD (i.e., warfarin)
* Current use of concomitant medications known to have adverse drug-drug interactions with CBD (i.e., valproate) or the potential to cause significant drug-drug interactions (i.e., clobazam).
* Known allergy to CBD or any ingredient of the study compound
* Currently enrolled in a clinical trial assessing the effects of an anti-pain intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ross, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data upon reasonable request. Requests should be directed to Stephen.ross@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were n=8 participants who were enrolled but failed screening/did not start the trial. Thus, the total number of participants who started the trial is n=6.
Period: Overall Study
Arm/Group | Cannabidiol (CBD) | Placebo (PCB)
Started | 5 | 1
Completed | 5 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cannabidiol (CBD) | Placebo (PCB) | Total
Number analyzed (Participants) | 5 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (10.533) | 54 (NA) — 1 participant - no standard deviation can be calculated. | 59.9 (10.533)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Opioid Analgesic Plasma Levels
Description: Opioid (i.e. the particular opioid used by a participant) analgesic plasma levels will be determined via High Performance Liquid Chromatography/Tandem Mass Spectrometry (LC-MS/MS).
Time Frame: Baseline, Week 2 Post-Initiation of Treatment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cannabidiol (CBD) | Placebo (PCB)
Number analyzed (Participants) | 5 | 1
ng/mL | 10.86 (14.35) | -11.4 (NA) — 1 Participant - standard deviation cannot be calculated.

2. Primary Outcome: Change in CBD Plasma Levels
Description: CBD plasma levels will be determined via High Performance Liquid Chromatography/Tandem Mass Spectrometry (LC-MS/MS).
Time Frame: Day 1 Post-Initiation of Treatment, Week 2 Post-Initiation of Treatment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cannabidiol (CBD) | Placebo (PCB)
Number analyzed (Participants) | 5 | 1
ng/mL | 38.28 (31.44) | 0 (NA) — 1 Participant - standard deviation cannot be calculated.

3. Secondary Outcome: Change in Score on Pain Catastrophizing Scale (PCS)
Description: PCS consists of 13 statements describing different thoughts and feelings that may be associated with pain. The degree to which one has these thoughts and feelings when experiencing pain is indicated on a scale of 0 (not at all) to 4 (all the time). The total range of score is 0-52, with a higher score indicating more frequent negative thoughts.
Time Frame: Baseline, Week 2 Post-Initiation of Treatment
Population: The participant in the Placebo (PCB) arm did not complete the PCS questionnaire at the Week 2 timepoint so change data was not collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol (CBD) | Placebo (PCB)
Number analyzed (Participants) | 5 | 0
score on a scale | 0.6 (8.65) |

4. Secondary Outcome: Change in Brief Pain Inventory (BPI) Score
Description: BPI - Short Form is a self-administered questionnaire. It evaluates:
  1. Pain intensity: 4 questions answered on a Likert scale of 0 (no pain) to 10 (pain as bad as you can imagine).
  2. Pain-related interference: 7 categories answered on a Likert scale of 0 (does not interfere) to 10 (completely interferes).
  The composite mean of these scores is used as the total pain interference score: the total score ranges from 0-55; higher scores indicate greater pain interference.
Time Frame: Baseline, Week 2 Post-Initiation of Treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol (CBD) | Placebo (PCB)
Number analyzed (Participants) | 5 | 0
score on a scale | -1.52 (1.49) |

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Safety and toxicity monitoring will be performed throughout the study for all participants. Safety variables to be assessed include AEs, vital signs, and safety laboratory values, when collected.
Arm/Group | Cannabidiol (CBD) | Placebo (PCB)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/1
Other Adverse Events (participants affected / at risk) | 5/5 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cannabidiol (CBD) (N=5) | Placebo (PCB) (N=1)
Left nephrolithiasis/pyelonephritis (requiring hospitalization) (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cannabidiol (CBD) (N=5) | Placebo (PCB) (N=1)
Urinary Tract Infection (Renal and urinary disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Left flank pain due to kidney stone (Renal and urinary disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1
Abnormal EKG (Cardiac disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 1
Bruise at IV site (Injury, poisoning and procedural complications) | 3 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Hypoalbuminemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Opiate Withdrawal (Psychiatric disorders) | 0 | 1
Heart Palpitations (Cardiac disorders) | 0 | 1
Somnolence (Nervous system disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Interrupted Sleep (Nervous system disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0
Bruise at IV Site (Injury, poisoning and procedural complications) | 3 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Imbalance (Nervous system disorders) | 1 | 0
Lightheadedness (Nervous system disorders) | 2 | 0
Hypotension (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Loose Stool (Gastrointestinal disorders) | 1 | 0
Pain at IV site (Injury, poisoning and procedural complications) | 1 | 0
Increased urination frequency (Renal and urinary disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Cardiac disorders) | 2 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT04760613/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT04760613/ICF_000.pdf